CLINICAL TRIAL: NCT04053413
Title: Pilot Study to Assess the Effectiveness of a Decision Tool for Cesarean Delivery vs. Trial of Labor
Brief Title: University of North Carolina-Healthwise Partnership Project on Birth Options Decision Aid
Acronym: B-READY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Healthwise (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-2023
Record Dates: First submitted 2019-08-05; First posted 2019-08-12 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Scar; Previous Cesarean Section; Vaginal Birth After Cesarean; Decision Making, Shared
MeSH Terms: conditions — Cicatrix | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Women in this group will undergo usual care and the complete the survey questions on knowledge and involvement in the decision for trial of labor after cesarean (TOLAC) or repeat cesarean.
- Decision Aid (Active Comparator): Women in this group will receive a decision aid prior to undergoing counseling by their physician. Following completion of the decision aid and physician counseling, they will complete a series of survey questions to assess their perceptions of their knowledge and involvement in the decision for trial of labor after cesarean (TOLAC) or repeat cesarean delivery.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — The decision aid is a series of web pages that includes videos, questions, and evidence-based information. The decision aid is designed to help women think about what matters to them and what questions they may have for their doctor or midwife. At the end, they receive a summary of which way they are leaning and what matters most to them.
  Arms: Decision Aid

SUMMARY:
This is pilot quasi-experimental study of women with one or two prior cesarean deliveries who are now pregnant and eligible for a trial of labor after cesarean delivery, to assess whether a decision aid, providing knowledge about trial of labor (VBAC) and planned repeat cesarean delivery can improve the birth options decision-making process for patients.

Participants are screened for eligibility through electronic health records. Once an individual is screened eligible, and email invite is sent providing information about the study and assessing the interest in participation. An on-line consent is completed and women are entered sequentially into the usual care group and then through further recruitment, another sample of women are entered into the decision aid group. The primary outcome is satisfaction with the shared decision-making process with their provider.

DETAILED DESCRIPTION:
Once a potential participant is screened eligible, completes the on-line informed consent, they are officially enrolled in the study and sent a link confirming their enrollment and the study group in which they have been assigned. Participants are sequentially enrolled in the study with enrollment first into the usual care group. Once enrollment in the usual care group is complete, enrollment into the decision aid group will occur.

The study includes two non-randomized groups:

Arm 1 (Usual care group): Women in this group will undergo usual care and complete the survey questions on knowledge of risks and benefits of TOLAC (also referred to as VBAC) and planned repeat cesarean (PRCS), certainty of their decision, and involvement in the decision for trial of labor (TOLAC) or repeat cesarean delivery.

Arm 2: (Decision aid group- group receiving the decision tool): Women in this group will receive a decision aid prior to undergoing counseling by their physician. Following completion of the decision aid and physician counseling, they will complete a series of survey questions to assess their knowledge of the risks and benefits of TOLAC and PRCS, certainty of their decision, and involvement in the decision for repeat cesarean or TOLAC.

The decision aid group will be compared with women who do not receive the decision aid (usual care group).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 19/0 and 36/6 weeks
* History of 1 or 2 prior cesarean deliveries

Exclusion Criteria:

* No contraindications to trial of labor after cesarean (TOLAC)
* No history of prior TOLAC

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Shared Decision Making (SDM) Process score | Up to 6 months prior to delivery
  This is a measure of the patient's involvement in the decision. 1 point is assigned for discussing the pros 'a lot' or 'some'; 1 point is assigned for discussing the cons 'a lot' or 'some'; 1 point is assigned for responding 'yes' if the provider explained the options; and 1 point is assigned for responding 'yes' that the provider asked the patient what treatment she wanted. The tool's score range is 0-4. A higher score indicates more involvement in the decision.

SECONDARY OUTCOMES:
Number of Participants (by category) With the Intent to Deliver by Repeat Cesarean Section or by Vaginal Delivery | Date of Admission
  Intended mode of delivery (repeat cesarean or vaginal) prior to actual delivery
Number of Participants (by category) who Delivered by Repeat Cesarean or Vaginal Delivery | Up to 72 hours after delivery
  Actual method of delivery (repeat cesarean or vaginal delivery)
Maternal or Fetal Complications at Delivery | Up to 72 hours after delivery
  Number of complication events: maternal postpartum hemorrhage, infection, fetal admission to neonatal intensive care unit.
Number of Participants (by Category) who desired Repeat Cesarean, Vaginal Delivery or Are Undecided after completion of the study survey | Up to 6 months prior to delivery
  Participant responses are: 1) repeat cesarean delivery, 2) vaginal delivery and 3) undecided

CONTACTS AND LOCATIONS:
Overall Officials: Wanda K Nicholson, MD, Principal Investigator — Univerisity of North Carolina - Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available 9 to 36 months following publication of the data as indicated in the section on Plan Description outlined above.
Access Criteria: Researchers will respond to letter or email requests from researchers with the plan description outlined in this section.
URL: https://research.unc.edu/clinical-trials/clinical-trials-gov/data-sharing-guidance/)

REFERENCES:
- [Derived] Venkatesh KK, Brodney S, Barry MJ, Jackson J, Lyons KM, Talati AN, Ivester TS, Munoz MC, Thorp JM, Nicholson WK. Patient decision aid for trial of labor after cesarean (TOLAC) versus planned repeat cesarean delivery: a quasi-experimental pre-post study. BMC Pregnancy Childbirth. 2021 Sep 23;21(1):650. doi: 10.1186/s12884-021-04119-3. PMID 34556061